CLINICAL TRIAL: NCT05561127
Title: Paclitaxel Coated Balloon for the Treatment of Chronic bEnigN sTricture- Bowel
Acronym: PATENT-B
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GIE Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR2053
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Bowel; Stricture
Keywords: dcb; bowel stricture; drug coated balloon; paclitaxel coated balloon
MeSH Terms: conditions — Constriction, Pathologic; Color Vision Defects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- GIE Medical ProTractX3 TTS DCB (Experimental): The ProTractX3 Drug-coated balloon is a 0.035" guidewire compatible over-the-wire catheter.
  Interventions: Combination Product: GIE Medical ProTractX3 TTS DCB
- Control (Active Comparator): Standard of Care.
  Interventions: Other: Control

INTERVENTIONS:
Combination Product: GIE Medical ProTractX3 TTS DCB — The ProTractX3 Drug-coated balloon is a 0.035" guidewire compatible over-the-wire catheter.
  Arms: GIE Medical ProTractX3 TTS DCB
Other: Control — Standard of Care Endoscopic Dilation
  Arms: Control

SUMMARY:
To determine the safety and efficacy of GIE Medical's ProTractX3™ TTS DCB for the treatment of recurrent benign bowel strictures.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 22
2. Diagnosis of symptomatic benign bowel stricture with at least 2 previous dilations.
3. Willing and able to complete protocol required follow up
4. Willing and able to provide written informed consent
5. Stricture length ≤ 5 cm

Exclusion Criteria:

1. Female subjects who are pregnant or breastfeeding or plan to get pregnant in next 12 months
2. Contraindication to endoscopy, anesthesia, or deep sedation.
3. Suspicion of malignant bowel stricture NOTE: Biopsy should be taken for every stricture during the initial endoscopy, however endoscopic balloon dilation may proceed without awaiting results if suspicion for malignancy is low in the opinion of the investigator.
4. Benign stricture due to extrinsic compression
5. Stricture is not amenable to standard balloon dilation (e.g. severe angulation, unable to pass guidewire, etc.)
6. Stricture complicated with abscess, fistula, perforation, leakage or varices
7. Stricture segment has moderate to severe active inflammation at the time of treatment. Moderate to severe inflammation is defined as any one of; ulcers >0.5cm in diameter, ulcerated surface >10%, affected (inflamed) surface >50%, marked erythema, absent vascular pattern, significant friability, or erosions
8. Multiple clinically significant strictures unable to be treated with a single balloon (i.e. total segment length must be ≤5cm) NOTE: Clinically significant strictures include those that are unable to be passed by the endoscope.
9. Received steroid injections into target stricture in the last 8 weeks
10. Stricture is not able to be dilated to ≥15mm in small bowel or ≥18mm in large bowel
11. Diagnosis of metastatic cancer of any type that is not considered in remission or non-metastatic cancer that may require radiation treatment in the pelvic region (e.g. prostate cancer)
12. Suspected perforation of gastrointestinal tract
13. Active systemic infection
14. Allergy to paclitaxel
15. Severe coagulation disorders or current use of anticoagulant or antiplatelet medication that cannot be safely managed per relevant societal guidelines
16. Chronic systemic steroid use (defined as greater than 10 mg/day) for any medical conditions unless subject is willing to undergo a 4-week washout and discontinue steroid use
17. Condition requiring treatment in urgent setting
18. Life expectancy of less than 24 months
19. Concurrent medical condition that would affect the investigator's ability to evaluate the patient's condition or could compromise patient safety, such as recent myocardial infarction, severe pulmonary disease, bleeding diathesis, large thoracic aneurysm, pharyngeal or cervical deformity, etc.
20. Current participation in another pre-market drug or medical device clinical study unless in long term follow-up

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from Stricture Recurrence | 6 Months Post-Treatment
  Endoscopic Obstruction Scale (EOS) of > 1 when using a pediatric colonoscope or equivalent
Primary Safety Outcome | 30 Days Post-Treatment
  Incidence of device- and/or procedure-related Major Adverse Events (MAEs) (Death, perforation of the esophagus, bleeding requiring intervention or transfusion)

SECONDARY OUTCOMES:
Freedom from clinically driven target stricture reintervention | 6 Months Post-Procedure
  Freedom from clinically driven reintervention represents freedom from repeat dilation, incision, or surgical management of the target stricture for recurrent obstructive symptoms.
Improvement in GIQLI-10 score | 6 Months Post-Procedure
  The Gastrointestinal Quality of Life Index (GIQLI) is a validated questionnaire developed as a health-related quality of life assessment tool for patients with gastrointestinal diseases. The items on the GIQLI-10 align closely with common obstructive symptoms found in patients with bowel strictures.

OTHER OUTCOMES:
Surgery Free Survival | 30 days, 3 months, 6 months, 12 months, and annually thereafter through 5 years
Improvement in GIQLI-10 | 30 days, 3 months, 6 months, 12 months, and annually thereafter through 5 years
Technical Success | 30 days, 3 months, 6 months, 12 months, and annually thereafter through 5 years
Improvement in EOS | 30 days, 3 months, 6 months, 12 months, and annually thereafter through 5 years
Dilations per year before and after treatment | 30 days, 3 months, 6 months, 12 months, and annually thereafter through 5 years
Time between dilations | 30 days, 3 months, 6 months, 12 months, and annually thereafter through 5 years
Estimated stricture diameter | 30 days, 3 months, 6 months, 12 months, and annually thereafter through 5 years

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Honor Health, Scottsdale, Arizona
  - University of California, Irvine, Irvine, California
  - Gastro Care Institute, Lancaster, California
  - Cedars Sinai, Los Angeles, California
  - San Diego Gastroenterology, San Diego, California
  - University of Colorado Anschutz, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Borland-Groover, Jacksonville, Florida
  - Research Associates of South Florida, Miami, Florida
  - Hillcrest Medical Research, Orange City, Florida
  - Orlando Health, Orlando, Florida
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Rush University, Chicago, Illinois
  - Kansas Gastroenterology, LLC, Wichita, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tandem Clinical Research, Marrero, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Rutgers University, Piscataway, New Jersey
  - New York Presbyterian Hospital- Columbia University Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor St. Luke's Medical Center, Houston, Texas
  - The University of Utah, Salt Lake City, Utah
  - Virginia Mason, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided